CLINICAL TRIAL: NCT00741676
Title: Comparison of the Laparoscopy-Assisted Distal Gastrectomy(LADG) and Open Distal Gastrectomy (ODG) for Advanced Gastric Cancer (Stage Ib and II).
Brief Title: Comparison of the Laparoscopy-Assisted Distal Gastrectomy and Open Distal Gastrectomy for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Institutional review board of Holy Family Hospital.The Catholic University of Korea, Department of Surgery.Holy Family Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HFHGS01
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-08

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Procedure: open distal gastrectomy
- 1 (Experimental)
  Interventions: Procedure: laparoscopy-assisted distal gastrectomy

INTERVENTIONS:
Procedure: laparoscopy-assisted distal gastrectomy — 10 mm trocar under umbilicus, 12 mm and 5 mm trocar at the right flank area are inserted into abdominal wall. Another two 5 mm trocar are inserted into the both midline of subcostal line. The devices for operation are inserted through the trocars. Subtotal gastrectomy (dissect more than 2/3 of stomach and total omentectomy) and D2 lymph node dissection (around common hepatic artery, celiac artery, proximal part of splenic artery, hepatoduodenal ligament, superior mesenteric vein) will be performed basically. As a general rule, Billroth II method was used for gastric reconstruction for all cases.Dissected stomach and lymph node are collected through additional 3~5 cm incision at the preexisting epigastric incision.Finally, Billroth II reconstruction is performed.
  Other Names: LADG
  Arms: 1
Procedure: open distal gastrectomy — Approximately 15~20 cm length incision is made from falciform process to periumbilical area. Subtotal gastrectomy (dissect more than 2/3 of stomach and total omentectomy) and D2 lymph node dissection (around common hepatic artery, celiac artery, proximal part of splenic artery, hepatoduodenal ligament, superior mesenteric vein) will be performed basically. As a general rule, Billroth II method was used for gastric reconstruction for all cases.
  Other Names: ODG
  Arms: 2

SUMMARY:
Among surgical methods for gastric cancer, incision about 15 ~20 cm length is prepared for open gastric cancer surgery while 0.5 ~ 1.2 cm is for laparoscopy gastric cancer surgery. Complications such as pain, abdominal adhesion, and problems associated with delayed recovery are common in open surgery because of large incision; however, those complications are less common in laparoscopy surgery because small sized incision is prepared. Range of surgery for curative dissection depends on the level of progress of a cancer, i.e., depends on whether gastric wall invasion, lymph node metastasis, or invasion to adjacent organs presented. Since recurrence in the lymph nodes after the operation is very common, the most important step in the gastric surgery is to dissect lymph node completely. According to the gastric cancer surgery manual published by Japan Gastric Cancer Association, more than D2 lymph node dissection is essential for improving survival rate in advanced gastric cancer. More than D2 lymph node dissection is relatively safely conducted by open surgery, whereas it is controversial in laparoscopy surgery because it is very hard to maintain surgical field under laparoscopic condition. Recently, widened rage of lymph node dissection by using laparoscopy is possible as laparoscopic surgical techniques are accumulated and new surgical devices are introduced. According to the case reports, D2 lymph node dissection by laparoscopy surgery shows similar results to the one by open surgery in aspects of recurrence rate and the number of dissected lymph node. Also, according to Hur and el., in case of upper gastric cancer, laparoscopy surgery is more useful to dissect #10 and #11 lymph node.In our prospective case study, the investigators would like to compare effectiveness, complications, patterns of recurrence, and survival rate between the two surgical approaches, laparoscopy distal gastrectomy and open distal gastrectomy. The investigators randomly operate the advanced gastric cancer patients, who need distal gastrectomy and D2 lymph node dissection. Surgical methods are selected randomly whether open surgery or laparoscopy surgery. Finally, the investigators wish our case report to contribute to the establishment of the safety and the effectiveness of laparoscopy surgery conducted for advanced gastric cancers. Consequently, our case report will contribute to establish the ideal surgical method for the advanced gastric cancer patients.

DETAILED DESCRIPTION:
In both arms,subtotal gastrectomy (dissect more than 2/3 of stomach and total omentectomy) and D2 lymph node dissection (around common hepatic artery, celiac artery, proximal part of splenic artery (4d, 4sb), hepatoduodenal ligament, superior mesenteric vein) wiil be performed basically. As a general rule, Billroth II method will be used for gastric reconstruction for all cases.Billroth II gastrectomy is to link the gastric pouch to the jejunum 10~15 cm distal to the ligament of Treitz. An antecolic or retrocolic gastrojejunostomy connects the jejunum to the stomach in one continuous segment. For anastomosis, absorbable suture is used. Anastomotic diameter is 5~6 cm length. Drainage tube is inserted through the right flank area and additional drainage tubes can be inserted as needed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic finding by gastric endoscopy: confirmed gastric adenocarcinoma
* Age: older than 20 year old, younger than 80 year old
* Cancer core: located at the middle or lower part of stomach
* Preoperative cancer stage (CT, GFS stage): cT2N0M0, cT2aN1M0, cT2bN1M0, cT3N0M0
* ASA score: ≤ 3
* Informed consent patients (explanation about our clinical trials is provided to the patients or patrons, if patient is not available)

Exclusion Criteria:

* Concurrent cancer patients or patient who was treated due to other types of cancer before the patient was diagnosed as a gastric cancer patient
* Patient who was treated by other types of treatment methods, such as chemotherapy, immunotherapy, or radiotherapy
* Patient who was received upper abdominal surgery (except, laparoscopic cholecystectomy)
* Patient who was treated because of systemic inflammatory disease
* Pregnant patient
* Patient who suffer from bleeding tendency disease, such as hemophilia or patient taking anti-coagulant medication due to deep vein thrombosis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
2 year survival | two year

SECONDARY OUTCOMES:
efficacy and clinical out come | two year

CONTACTS AND LOCATIONS:
Overall Officials: Wook Kim, Professor, Study Chair — Department of Surgery, Holy Family Hospital. The Catholic University of Korea
Locations (2):
- South Korea (2):
  - Department of Surgery, Holy Family Hospital. College of Medicine. The Catholic University of Korea, Pucheon, Gyeonggi-do
  - Department of Surgery, Holy Family Hospital, The Catholic University of Korea, Bucheon-si, Gyunggi Do

REFERENCES:
- [Background] Yano H, Monden T, Kinuta M, Nakano Y, Tono T, Matsui S, Iwazawa T, Kanoh T, Katsushima S. The usefulness of laparoscopy-assisted distal gastrectomy in comparison with that of open distal gastrectomy for early gastric cancer. Gastric Cancer. 2001;4(2):93-7. doi: 10.1007/pl00011730. PMID 11706767
- [Background] Mochiki E, Kamiyama Y, Aihara R, Nakabayashi T, Asao T, Kuwano H. Laparoscopic assisted distal gastrectomy for early gastric cancer: Five years' experience. Surgery. 2005 Mar;137(3):317-22. doi: 10.1016/j.surg.2004.10.012. PMID 15746786
- [Background] Morita M, Baba H, Fukuda T, Taketomi A, Kohnoe S, Seo Y, Saito T, Tomoda H, Sugimachi K. Submucosal gastric cancer with lymph node metastasis. J Surg Oncol. 1998 May;68(1):5-10. doi: 10.1002/(sici)1096-9098(199805)68:13.0.co;2-b. PMID 9610656
- [Background] Nakajima T. Gastric cancer treatment guidelines in Japan. Gastric Cancer. 2002;5(1):1-5. doi: 10.1007/s101200200000. PMID 12021853
- [Background] Noshiro H, Nagai E, Shimizu S, Uchiyama A, Tanaka M. Laparoscopically assisted distal gastrectomy with standard radical lymph node dissection for gastric cancer. Surg Endosc. 2005 Dec;19(12):1592-6. doi: 10.1007/s00464-005-0175-9. Epub 2005 Oct 24. PMID 16247578
- [Background] Lee JH, Kim YW, Ryu KW, Lee JR, Kim CG, Choi IJ, Kook MC, Nam BH, Bae JM. A phase-II clinical trial of laparoscopy-assisted distal gastrectomy with D2 lymph node dissection for gastric cancer patients. Ann Surg Oncol. 2007 Nov;14(11):3148-53. doi: 10.1245/s10434-007-9446-0. Epub 2007 Aug 20. PMID 17705092
- [Background] Ageno W, Squizzato A, Garcia D, Imberti D. Epidemiology and risk factors of venous thromboembolism. Semin Thromb Hemost. 2006 Oct;32(7):651-8. doi: 10.1055/s-2006-951293. PMID 17024592
- [Background] Huscher CG, Mingoli A, Sgarzini G, Brachini G, Binda B, Di Paola M, Ponzano C. Totally laparoscopic total and subtotal gastrectomy with extended lymph node dissection for early and advanced gastric cancer: early and long-term results of a 100-patient series. Am J Surg. 2007 Dec;194(6):839-44; discussion 844. doi: 10.1016/j.amjsurg.2007.08.037. PMID 18005781
- [Background] Sasako M, Saka M, Fukagawa T, Katai H, Sano T. Surgical treatment of advanced gastric cancer: Japanese perspective. Dig Surg. 2007;24(2):101-7. doi: 10.1159/000101896. Epub 2007 Apr 19. PMID 17446702
- [Background] Song KY, Kim SN, Park CH. Laparoscopy-assisted distal gastrectomy with D2 lymph node dissection for gastric cancer: technical and oncologic aspects. Surg Endosc. 2008 Mar;22(3):655-9. doi: 10.1007/s00464-007-9431-5. PMID 17593447
- [Background] Kim MC, Kim KH, Kim HH, Jung GJ. Comparison of laparoscopy-assisted by conventional open distal gastrectomy and extraperigastric lymph node dissection in early gastric cancer. J Surg Oncol. 2005 Jul 1;91(1):90-4. doi: 10.1002/jso.20271. PMID 15999352
- [Background] Hur H, Jeon HM, Kim W. Laparoscopic pancreas- and spleen-preserving D2 lymph node dissection in advanced (cT2) upper-third gastric cancer. J Surg Oncol. 2008 Feb 1;97(2):169-72. doi: 10.1002/jso.20927. PMID 18095269
- [Derived] Lee J, Kim W. Long-term outcomes after laparoscopy-assisted gastrectomy for advanced gastric cancer: analysis of consecutive 106 experiences. J Surg Oncol. 2009 Dec 15;100(8):693-8. doi: 10.1002/jso.21400. PMID 19731245